CLINICAL TRIAL: NCT01591928
Title: Heterotaxy Syndrome and Intestinal Rotation Abnormalities - A Prospective Study
Status: Completed | Type: Observational
Sponsor: University of Alberta (Other)
Responsible Party: Principal Investigator, Lindsay Ryerson, Assistant Professor, University of Alberta
Other Study IDs: 2012-LR-01
Record Dates: First submitted 2012-05-02; First posted 2012-05-04 (Estimated); Last update posted 2018-12-19 (Actual); Status verified 2018-12

CONDITIONS: Heterotaxy Syndrome
Keywords: Pediatrics; Congenital heart disease; Heterotaxy syndrome; Intestinal malrotation
MeSH Terms: conditions — Heterotaxy Syndrome; Heart Defects, Congenital; Volvulus Of Midgut

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Infants with heterotaxy syndrome

SUMMARY:
Infants with heterotaxy syndrome (HS) are born with an abnormal arrangement of organs along the right-left body axis. Abnormalities of intestinal rotation and fixation are commonly associated with HS. Malrotation is the most worrisome intestinal rotation abnormality (IRA). Advances in cardiac surgery have improved HS mortality such that there is increasing attention to IRA and their management. The objective of this research project is to prospectively observe a cohort of infants with HS and IRA and evaluate their long term outcomes. Specifically, the investigators would like to determine what is the natural history of asymptomatic IRA in patients with HS and what is the morbidity and mortality secondary to an elective Ladd procedure for asymptomatic IRA in a population with HS? The investigators plan a prospective, multi-center, observational study to follow this complicated group of patients. This will be a web-based database collected from major cardiac tertiary care centers in both Canada and the United States. Patients with HS will be recruited by their primary site and clinical data will be collected by their primary site prospectively throughout childhood until they are at least five years of age. This patient population will be followed by their own clinical care givers; this is not an interventional study. No additional clinic visits will be required and the patients will not have to be contacted. Patient medical records will be accessed by a member of the study team at the primary site at least once per year or more frequently if interventions are required or complications develop.

ELIGIBILITY:
Inclusion Criteria:

* All infants less than or equal to six months of age with a new diagnosis of heterotaxy syndrome

Exclusion Criteria:

Ages: 1 Day to 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: All infants with heteterotaxy syndrome whose families provide written informed consent.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2012-03; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Midgut volvulus | First year of life
  Surgical intervention

SECONDARY OUTCOMES:
Morbidity secondary to a prophylactic Ladd procedure | Post Ladd procedure
Mortality secondary to a prophylactic Ladd procedure | Within one month of Ladd procedure

CONTACTS AND LOCATIONS:
Overall Officials: Lindsay Ryerson, MD, Principal Investigator — University of Alberta
Locations (1):
- Stollery Children's Hospital, Edmonton, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No